CLINICAL TRIAL: NCT02004613
Title: Ancillary Effects of Dexmedetomidine Sedation After Cardiac Surgery
Acronym: Decade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Alparslan Turan, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1379
Record Dates: First submitted 2013-08-01; First posted 2013-12-09 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine infusion, without a bolus dose, (or a comparable volume of placebo) will be initiated before the surgical incision at a rate of 0.1 mcg/kg/hr at the end of bypass, the dose will be increased to 0.2 mcg/kg/hr. Postoperatively patients will continue to receive the study medication at a rate of 0.4mcg/kg/hr. The study medication infusion will be continued for a total of 24 hours from the initial administration time intra-operatively.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): normal saline administration matching dexmedetomidine rate of infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Placebo — Normal saline administration matching dexmedetomidine rate of infusion
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Ancillary Effects of Dexmedetomidine Sedation After Cardiac Surgery

DETAILED DESCRIPTION:
The investigator goal is to evaluate the effects of intraoperative and postoperative dexmedetomidine sedation (versus placebo after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old;
2. Scheduled for cardiac surgery with bypass (CABG, valve, or combined);
3. Able to provide a written informed consent;
4. Hemodynamically stable (heart rate>= 55).

Exclusion Criteria:

1. Sick sinus syndrome or Wolff-Parkinson-White syndrome
2. Atrio-ventricular block
3. Hypersensitivity or known allergy to dexmedetomidine
4. Hepatic disease, e.g. twice the normal level of liver enzymes
5. Atrial fibrillation within 1 preoperative month;
6. Permanent pacemaker;
7. Use of amiodarone or dexmedetomidine within the last 30 days;
8. Patients with an ejection fraction under 30% or who had severe heart failure
9. Myocardial infarction in the previ¬ous 7 days;
10. Body mass index =< 40 (BMI= mass (kg) / height (m)2);
11. Those taking clonidine within last 48 hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — Staff member
Locations (1):
- Cleveland Clinic Main, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Turan A, Duncan A, Leung S, Karimi N, Fang J, Mao G, Hargrave J, Gillinov M, Trombetta C, Ayad S, Hassan M, Feider A, Howard-Quijano K, Ruetzler K, Sessler DI; DECADE Study Group. Dexmedetomidine for reduction of atrial fibrillation and delirium after cardiac surgery (DECADE): a randomised placebo-controlled trial. Lancet. 2020 Jul 18;396(10245):177-185. doi: 10.1016/S0140-6736(20)30631-0. PMID 32682483

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 400 | 398
Completed | 398 | 396
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 398 | 396 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only reported the mean and standard deviation for each group. Age is not available for 4 patients.
  years
    number analyzed (Participants) | 396 | 394 | 790
    (all) | 63 (11) | 62 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 4 patients sex data were not availiable.
  Participants
    number analyzed (Participants) | 396 | 394 | 790
    Female | 132 | 111 | 243
    Male | 264 | 283 | 547
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 5 patients didn't had availiable race data.
  Participants
    Race: number analyzed (Participants) | 395 | 394 | 789
    Race: white | 365 | 363 | 728
    Race: not white | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  United States | 398 | 396 | 794
Modified Brief Pain Inventory [Count of Participants; unit: Participants] — Population: 44 patients' baseline MBPI information was not available. Any overall severity means any pain in the last 24 hours. Any pain inference means any pain that interfering with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life in the last 24 hours.
  Participants
    Overall Severity (any): number analyzed (Participants) | 374 | 376 | 750
    Overall Severity (any) | 95 | 89 | 184
    Pain interference (any) | 85 | 83 | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Atrial Arrhythmia
Description: The occurrence of postoperative atrial arrhythmias
Time Frame: From the end of surgery to postoperative day 5
Population: 2 patients had no Atrial Arrhythmia data.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 397 | 395
Participants | 121 | 134
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Hypothesis: dexmedetomidine would reduce the incidence of postoperative atrial arrhythmias; Test type: Superiority; p = 0.34, Regression, Logistic; Risk Ratio (RR) = 0.91, 97.8% CI 2-sided [0.72 to 1.15]

2. Primary Outcome: Number of Patients With Delirium
Description: The occurrence of postoperative delirium
Time Frame: From the end of surgery to postoperative day 5
Population: Delirium data is not available in 18 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 389 | 387
Participants | 67 | 46
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; hypothesis: Dexmedetomidine may reduce the incidence of postoperative delirium; Test type: Superiority; p = 0.026, Regression, Logistic; Risk Ratio (RR) = 1.48, 97.8% CI 2-sided [0.99 to 2.23]

3. Secondary Outcome: Number of Patients With Acute Kidney Injury
Description: Acute kidney injury is defined according to Acute Kidney Injury Network (AKIN) classifications. No risk means no risk of acute kidney injury, while a higher stage means worse kidney function.
Time Frame: From the end of surgery to postoperative day 5
Population: Acute kidney injury data is not available in 16 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 389 | 389
Participants
  No risk | 348 | 359
  stage1 | 33 | 29
  Stage2 | 4 | 0
  Stage3 | 4 | 1
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Test type: Superiority; p = 0.14, Regression, Logistic; Risk Ratio (RR) = 1.40, 97.5% CI 2-sided [0.84 to 2.34]

4. Secondary Outcome: Number of Patients With Incisional Pain
Description: Patients were evaluated at 90 days by modified Brief Pain Inventory.
Time Frame: 90 days after surgery
Population: Incisional pain at 90 days is not available in 205 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 289 | 300
Participants | 79 | 93
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Test type: Other; p = 0.29, Regression, Logistic; Risk Ratio (RR) = 0.87, 97.5% CI 2-sided [0.65 to 1.16]

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/394 | 1/390
Serious Adverse Events (participants affected / at risk) | 21/394 | 8/390
Other Adverse Events (participants affected / at risk) | 234/394 | 154/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine (N=394) | Placebo (N=390)
Hemorrhage (Blood and lymphatic system disorders) | 4 | 3
asystol (Cardiac disorders) | 1 | 1
heart failure (Cardiac disorders) | 1 | 0
re-intervention (Cardiac disorders) | 0 | 1 — The patient went back to the operation room for redo complex mitral valve repair with plication
infection (Infections and infestations) | 2 | 0
seizure (Nervous system disorders) | 0 | 1
stroke (Nervous system disorders) | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 — Elevated troponin postoperatively
Pericardial effusion (Cardiac disorders) | 1 | 0
Transient Ischemic attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexmedetomidine (N=394) | Placebo (N=390)
Clinically important bradycardia (Cardiac disorders) | 36 | 45
Clinically important hypotension (Blood and lymphatic system disorders) | 224 | 140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02004613/Prot_SAP_000.pdf